CLINICAL TRIAL: NCT05489224
Title: A Randomized, Active-Controlled, Double-Blind, Phase 3 Study to Compare Efficacy and Safety of Two Intravenous Infusion Formulations of Tocilizumab (CT-P47 and RoActemra) When Co-administered With Methotrexate in Patients With Rheumatoid Arthritis
Brief Title: A Study to Compare Efficacy and Safety of CT-P47 and RoActemra in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P47 3.1
Record Dates: First submitted 2022-07-24; First posted 2022-08-05 (Actual); Results first posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P47 (Experimental): CT-P47(Tocilizumab)
  Interventions: Biological: CT-P47
- EU-approved RoActemra (Active Comparator): EU-approved RoActemra(Tocilizumab)
  Interventions: Biological: CT-P47; Biological: EU-approved RoActemra

INTERVENTIONS:
Biological: CT-P47 — CT-P47, 8 mg/kg (not exceeding 800 mg/dose) by intravenous (IV) infusion every 4 weeks (Q4W)
Biological: EU-approved RoActemra — EU-approved RoActemra, 8 mg/kg (not exceeding 800 mg/dose) by IV infusion Q4W
  Arms: EU-approved RoActemra

SUMMARY:
This is a phase 3 study to compare efficacy and safety of CT-P47 and RoActemra in patients with moderate to severe active rheumatoid arthritis.

DETAILED DESCRIPTION:
CT-P47, containing the active ingredient tocilizumab, is a recombinant humanized monoclonal antibody that is being developed as a similar biological medicinal product to RoActemra/Actemra. The purpose of this study is to demonstrate similar efficacy and safety of CT-P47 and RoActemra in patients with moderate to severe rheumatoid arthritis when co-administered with methotrexate.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is male or female aged 18 to 75 years old, both inclusive.
2. Patient has had a diagnosis of RA according to the 2010 ACR/EULAR classification criteria for at least 24 weeks prior to the first administration of the study drug.

Exclusion Criteria:

1. Patient who has previously received investigational or licensed product; targeted synthetic DMARD(s) (e.g., tofacitinib, baricitinib) for the treatment of RA and/or an interleukin-6 (IL-6) inhibitor for any purposes.
2. Patient who has previously received more than 1 biologic agents approved for the treatment of RA.
3. Patient who has allergies to any of the excipients of study drug or any other murine and human proteins, or patient with a hypersensitivity to immunoglobulin products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Klimiuk Piotr, Principal Investigator — INTER CLINIC Piotr Adrian Klimiuk
Locations (1):
- INTER CLINIC Piotr Adrian Klimiuk, Bialystok, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burmester G, Trefler J, Racewicz A, Jaworski J, Zielinska A, Krogulec M, Jeka S, Wojciechowski R, Kolossa K, Dudek A, Krajewska-Wlodarczyk M, Hrycaj P, Klimiuk PA, Kim S, Suh J, Yang G, Kim Y, Jung Y, Park G, Smolen JS. Efficacy and Safety of Biosimilar CT-P47 Versus Reference Tocilizumab: 1-Year Results of a Randomised, Active-Controlled, Double-Blind, Phase III Study in Patients with Rheumatoid Arthritis. Clin Drug Investig. 2025 Aug;45(8):551-563. doi: 10.1007/s40261-025-01453-8. Epub 2025 Jul 12. PMID 40650731

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P47/CT-P47 Maintenance: Treatment Period I: Patients who were initially randomly assigned to CT-P47 in Treatment Period I (from Week 0 to Week 20).
  Treatment Period II: All patients who received CT-P47 in Treatment Period I and continued to receive CT-P47 in Treatment Period II (from Week 24 to Week 48).
- RoActemra/RoActemra Maintenance: Treatment Period I: Patients who were initially randomly assigned to RoActemra in Treatment Period I (from Week 0 to Week 20).
  Treatment Period II: Patients who received RoActemra in Treatment Period I and re-randomized to continue RoActemra in Treatment Period II (from Week 24 to Week 48).
- Switched to CT-P47: Treatment Period I: Not applicable
  Treatment Period II: Patients who received RoActemra in Treatment Period I and re-randomized to receive CT-P47 in Treatment Period II (from Week 24 to Week 48).
Period: Treatment Period I
Arm/Group | CT-P47/CT-P47 Maintenance | RoActemra/RoActemra Maintenance | Switched to CT-P47
Started | 234 | 237 | 0
Completed (Patients who completed study drug administration in Treatment Period I) | 225 | 219 | 0
Not Completed | 9 | 18 | 0
Not completed — Withdrawal by Subject | 6 | 5 | 0
Not completed — Adverse Event | 3 | 11 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Period: Treatment Period II up to Week 32
Arm/Group | CT-P47/CT-P47 Maintenance | RoActemra/RoActemra Maintenance | Switched to CT-P47
Started (Patients who had administrated RoActemra during Treatment Period I has been re-randomized in a 1:1 ratio into 2 groups - RoActemra Maintenance and switched to CT-P47.) | 225 | 109 | 110
Completed (This data summary is based on the Week 32 results, so all patients were considered as Not Completed (whole study period; Week 52). All patients were considered as ongoing at the time of Week 32 data cut-off.) | 0 | 0 | 0
Not Completed | 225 | 109 | 110
Not completed — Ongoing | 222 | 107 | 107
Not completed — Adverse Event | 3 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- CT-P47: Patients who were initially randomly assigned to CT-P47 in Treatment Period I.
- RoActemra: Patients who were initially randomly assigned to RoActemra in Treatment Period I.
- Total: Total of all reporting groups
Arm/Group | CT-P47 | RoActemra | Total
Number analyzed (Participants) | 234 | 237 | 471
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (10.98) | 54.4 (11.61) | 54.8 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 180 | 361
  Male | 53 | 57 | 110
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 234 | 237 | 471
  Race: Other | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 6 | 4 | 10
  Ethnicity: Non-Hispanic or Non-Latino | 228 | 233 | 461
Body Weight on Day 1 [Count of Participants; unit: Participants]
  <100 kg | 208 | 210 | 418
  ≥100 kg | 26 | 27 | 53
DAS28 (ESR) score at Screening [Count of Participants; unit: Participants] — The DAS28(ESR) score was derived using the following formulae:
  DAS28 (ESR)=(0.56 ×√TJC28)+(0.28 × √SJC28)+(0.70 × ln[ESR])+(0.014 ×GH)
  Where:
  * TJC28 = number of tender joints (0-28): tender joint count (TJC)
  * SJC28 = number of swollen joints (0-28): swollen joint count (SJC)
  * ESR = ESR measurement (mm/hour)
  * GH = patient's global disease activity measured on 100 mm VAS
  DAS28 (ESR) >5.1 was condisered to be a higher disease activity than DAS28 (ESR) ≤5.1.
  Participants
    DAS28 (ESR) >5.1 | 229 | 230 | 459
    DAS28 (ESR) ≤5.1 | 5 | 7 | 12
Prior biologic use approved for RA treatment [Count of Participants; unit: Participants]
  Yes | 58 | 62 | 120
  No | 176 | 175 | 351

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Disease Activity Score 28 (DAS28) Using Erythrocyte Sedimentation Rate (ESR) at Week 24
Description: The DAS28(ESR) score was derived using the following formulae:
  DAS28 (ESR)=(0.56 ×√TJC28)+(0.28 × √SJC28)+(0.70 × ln[ESR])+(0.014 ×GH)
  Where:
  * TJC28 = number of tender joints (0-28): tender joint count (TJC)
  * SJC28 = number of swollen joints (0-28): swollen joint count (SJC)
  * ESR = ESR measurement (mm/hour)
  * GH = patient's global disease activity measured on VAS (mm: 0-100)
  DAS28 (ESR) values could be ranged from 0 to 10 while higher values mean a higher disease activity.
Time Frame: Week 24
Population: ITT set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | CT-P47 | RoActemra
Number analyzed (Participants) | 234 | 237
units on a scale | -3.77 (0.120) | -3.67 (0.118)
Statistical Analysis 1: Comparison: CT-P47 vs RoActemra; Test type: Equivalence — Predefined margin: -0.6 to 0.5; ANCOVA; ANCOVA with multiple imputation; Treatment difference and 90% CI = -0.10, 90% CI 2-sided [-0.30 to 0.10]

2. Secondary Outcome: Mean Change From Baseline in DAS28 (ESR) at Week 32
Description: as for outcome 1
Time Frame: Week 32
Population: ITT-Treatment Period II Subset
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CT-P47 Maintenance: Patients who received CT-P47 during Treatment Period I and continued to receive CT-P47 in Treatment Period II.
- RoActemra Maintenance: Patients who were initially randomly assigned to RoActemra at Day 1 (Week 0) and re-randomized (1:1 ratio) at Week 24 to continue to receive RoActemra in Treatment Period II.
- Switched to CT-P47: Patients who were initially randomly assigned to RoActemra at Day 1 (Week 0) and re-randomized (1:1 ratio) at Week 24 to undergo transition to CT-P47 in Treatment Period II.
Arm/Group | CT-P47 Maintenance | RoActemra Maintenance | Switched to CT-P47
Number analyzed (Participants) | 225 | 109 | 110
units on a scale | -3.921 (1.2548) | -3.994 (1.1753) | -4.218 (1.1380)

3. Secondary Outcome: ACR20, ACR50, and ACR70 Response Rate at Week 24
Description: ACR20 is defined as both improvement of 20% in the number of tender and number of swollen joints, and a 20% improvement in the three of the following five criteria: 1) patient global assessment of disease activity, 2) physician global assessment of disease activity, 3) functional ability measure using Health Assessment Questionnaire (HAQ), 4) visual analog pain scale, and 5) erythrocyte sedimentation rate (ESR) or C-reactive protein (CRP). ACR50 and ACR70 are the same instruments with improvement levels defined as 50% and 70% respectively versus 20% for ACR20.
Time Frame: Week 24
Population: ITT set
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P47 | RoActemra
Number analyzed (Participants) | 234 | 237
Participants
  ACR20 | 199 | 189
  ACR50 | 142 | 146
  ACR70 | 100 | 99

4. Secondary Outcome: ACR20, ACR50, and ACR70 Response Rate at Week 32
Description: as for outcome 3
Time Frame: Week 32
Population: ITT-Treatment Period II Subset
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P47 Maintenance | RoActemra Maintenance | Switched to CT-P47
Number analyzed (Participants) | 225 | 109 | 110
Participants
  ACR20 | 199 | 96 | 98
  ACR50 | 148 | 79 | 77
  ACR70 | 91 | 47 | 61

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from the date the patient signed the Informed Consent Form (ICF) until 4 weeks after the last study drug administration (up to 52 weeks [End-of-study visit]). For Treatment Period II in this page, results up to Week 32 cut-off of the first CSR were included.
Description: Treatment Period I: From Week 0 to prior to the 1st dosing in Treatment Period II. TEAEs with an actual/imputed start date prior to the 1st dosing in Treatment Period II, or TEAEs for those patients who did not administer study drug during Treatment Period II were included.
  Treatment Period II: From the 1st dosing in Treatment Period II to Week 32. TEAEs with an actual/imputed start date on or after the date of 1st dosing in Treatment Period II were included.
Groups:
- Treatment Period I: CT-P47: Patients who were initially randomly assigned to CT-P47 in Treatment Period I
- Treatment Period I: RoActemra: Patients who were initially randomly assigned to RoActemra in Treatment Period I
- Treatment Period II: CT-P47 Maintenance: Patients who received CT-P47 during Treatment Period I and continued to receive CT-P47 in Treatment Period II
- Treatment Period II: RoActemra Maintenance: Patients who were initially randomly assigned to RoActemra at Day 1 (Week 0) and re-randomized (1:1 ratio) at Week 24 to continue to receive RoActemra in Treatment Period II
- Treatment Period II: Switched to CT-P47: Patients who were initially randomly assigned to RoActemra at Day 1 (Week 0) and re-randomized (1:1 ratio) at Week 24 to undergo transition to CT-P47 in Treatment Period II
Arm/Group | Treatment Period I: CT-P47 | Treatment Period I: RoActemra | Treatment Period II: CT-P47 Maintenance | Treatment Period II: RoActemra Maintenance | Treatment Period II: Switched to CT-P47
All-Cause Mortality (participants affected / at risk) | 0/234 | 0/237 | 1/225 | 0/109 | 0/110
Serious Adverse Events (participants affected / at risk) | 10/234 | 9/237 | 4/225 | 3/109 | 2/110
Other Adverse Events (participants affected / at risk) | 140/234 | 143/237 | 54/225 | 26/109 | 23/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period I: CT-P47 (N=234) | Treatment Period I: RoActemra (N=237) | Treatment Period II: CT-P47 Maintenance (N=225) | Treatment Period II: RoActemra Maintenance (N=109) | Treatment Period II: Switched to CT-P47 (N=110)
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Lyme disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Peritonitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Bone loss (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Interferon gamma release assay positive (Investigations) | 0 | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Cervical cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Period I: CT-P47 (N=234) | Treatment Period I: RoActemra (N=237) | Treatment Period II: CT-P47 Maintenance (N=225) | Treatment Period II: RoActemra Maintenance (N=109) | Treatment Period II: Switched to CT-P47 (N=110)
Leukopenia (Blood and lymphatic system disorders) | 20 | 25 | 11 | 0 | 7
Lymphopenia (Blood and lymphatic system disorders) | 9 | 13 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 19 | 23 | 5 | 2 | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 8 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 3 | 8 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 18 | 19 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 9 | 4 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 50 | 40 | 10 | 7 | 4
Latent tuberculosis (Infections and infestations) | 0 | 0 | 12 | 2 | 3
Alanine aminotransferase increased (Investigations) | 37 | 48 | 17 | 7 | 5
Aspartate aminotransferase increased (Investigations) | 12 | 17 | 10 | 5 | 5
Transaminases increased (Investigations) | 6 | 11 | 0 | 0 | 0
Blood creatine phosphokinase MB increased (Investigations) | 0 | 0 | 5 | 5 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 16 | 19 | 0 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 8 | 5 | 0 | 0 | 0
Headache (Nervous system disorders) | 7 | 9 | 0 | 0 | 0
Hypertension (Vascular disorders) | 9 | 12 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT05489224/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT05489224/SAP_001.pdf